CLINICAL TRIAL: NCT04002635
Title: Endometrial Preparation Using Letrozole Compared to Artificial Cycle for Frozen Embryo Transfer in PCOS Patients
Brief Title: Letrozole for Frozen Embryo Transfer (FET) in Patients With Polycystic Ovary Syndrome (PCOS)
Acronym: LEFT
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Practical issues
Sponsor: CRG UZ Brussel (Other)
Collaborators: University Hospital, Ghent (Other)
Responsible Party: Principal Investigator, Liese Boudry, Medical doctor, CRG UZ Brussel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019LEFT001
Record Dates: First submitted 2019-06-27; First posted 2019-06-28 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Infertility, Female; Polycystic Ovary Syndrome; IVF; Ovulation Disorder
Keywords: frozen embryo transfer
MeSH Terms: conditions — Infertility, Female; Polycystic Ovary Syndrome | interventions — Letrozole; Estradiol; Progesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hormonal Replacement Therapy (Active Comparator): Artificial preparation of the endometrium using estradiol valerate 2mg 3x/day, and vaginal micronized progesterone 2x 400mg/day.
  Interventions: Drug: estradiol valerate
- Letrozole (Experimental): Using letrozole for ovulation induction before planning the frozen embryo transfer
  Interventions: Drug: Letrozole

INTERVENTIONS:
Drug: Letrozole — Letrozole ovulation induction
  Arms: Letrozole
Drug: estradiol valerate — hormonal replacement therapy
  Other Names: progesterone
  Arms: Hormonal Replacement Therapy

SUMMARY:
To offer patients with oligomenorrhoea or amenorrhoea an alternative to frozen embryo transfer in an artificial cycle, endometrial preparation using letrozole may be a valuable option. Letrozole, a potent, reversible nonsteroidal aromatase inhibitor with relatively short half-life, can successfully induce ovulation without any adverse anti-estrogenic effects and thus without affecting the endometrium. The use of letrozole typically results in monofollicular growth and this reduces the effect of supraphysiological levels of estrogen on the endometrium and embryo. The purpose of this study is to compare a frozen-thawed embryo transfer in an artificial cycle with a letrozole-induced ovulatory cycle, specifically in PCOS patients. The primary outcome is early pregnancy loss.

ELIGIBILITY:
Inclusion Criteria:

* Age more than or equal to 18 and less than or equal to 40
* BMI more than or equal to 18 and less than or equal to 35
* Diagnosis of PCOS according to Rotterdam criteria
* Normal gynaecological ultrasound < 6 months before inclusion
* Signed informed consent form
* Day 5 or 6 frozen-thawed embryo transfer, blastocyst stage

Exclusion Criteria:

* Recurrent implantation failure
* Recurrent miscarriage
* Presence of adenomyosis
* Untreated intrauterine pathology
* rAFS (revised American Fertility Society) Grade III or IV endometriosis
* Hydrosalpinx
* In vitro maturation (IVM)
* Untreated autoimmune disorders
* (History of) malignancy
* Allergy or reaction to the use of progynova, utrogestan and/or letrozole in the past
* Pre-implantation genetic testing (PGT)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-04-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
early pregnancy loss | 12 weeks after frozen embryo transfer

SECONDARY OUTCOMES:
cancellation rate | 2 months
number of visits to the clinic | 2 months
endometrial thickness on the day of planning of FET | 1 day
implantation rate | 1 day
biochemical and clinical pregnancy rate | 12 weeks
live birth rate | 1 year
neonatal birth weight | 1 year
term of delivery | 1 year
hypertensive disorders of pregnancy | 1 year

IPD SHARING:
Plan to Share IPD: Yes
Sharing with other study site, UZ Gent
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code